CLINICAL TRIAL: NCT01600859
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Oral Doses of E2609 in Subjects With Mild Cognitive Impairment or Mild Dementia Due to Alzheimer's Disease
Brief Title: Evaluation of E2609 in Subjects With Mild Cognitive Impairment or Mild Dementia Due to Alzheimer's Disease (Study: E2609-A001-101 Amendment 02)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E2609-A001-101
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- E2609 (Experimental)
  Interventions: Drug: E2609
- Placebo for E2609 (Placebo Comparator)
  Interventions: Drug: Placebo for E2609

INTERVENTIONS:
Drug: E2609 — E2609 capsules: 5 mg, 25 mg, 50 mg, and 200 mg
  E2609 doses: 5 mg, 10 mg, 25 mg, 50 mg, 100 mg, 200 mg, and 400 mg
  According to the randomized study design, participants who are assigned to receive E2609 will each receive a single assigned dose consisting of two capsules of E2609 or in some cases one capsule of E2609 and one of placebo
  Arms: E2609
Drug: Placebo for E2609 — Placebo capsules
  According to the randomized study design, participants who are assigned to receive placebo will each receive a single dose consisting of two capsules of placebo
  Arms: Placebo for E2609

SUMMARY:
Subjects will be adults aged 50 to 85 years who have subjective memory complaints and mild cognitive impairment or mild dementia due to Alzheimer's disease (AD). Subjects taking thyroxine or thyroid supplements and subjects receiving an acetylcholinesterase inhibitor (AChEI) and/or memantine for AD must be on a stable dose for at least 12 weeks prior to Screening and remain on their stable dose throughout the trial. Subjects will receive placebo or a single oral dose of E2609. Safety assessments will be conducted. Additionally, the pharmacokinetics of E2609 and drug effects will be evaluated using cerebrospinal fluid biomarkers and cognitive and psychological measures.

ELIGIBILITY:
Inclusion criteria:

* Meets the current cognitive classification of MCI or mild dementia due to AD pathology (all subjects having a "positive" biomarker for amyloid β) as defined by the National Institute on Aging - Alzheimer's Association (NIA-AA) research criteria
* Aged 50 to 85 years, inclusive at time of consent

Exclusion criteria:

* Currently has any neurological condition other than AD (Alzheimer's disease)-related that could be contributing to the subject's cognitive impairment
* Significant pathological findings on brain MRI at Screening, including but not limited to multiple microhemorrhages
* Any psychiatric diagnosis or symptoms, e.g., hallucinations, major depression,anxiety or delusions that in the Investigator's opinion could interfere with assessment of cognition or confound the diagnosis of MCI or mild dementia due to AD in the subject.
* A lifetime history of cerebrovascular events or non-vasovagal related loss of consciousness within the last 10 years
* Any other abnormality of the ECG at Screening and/or Baseline (including QRS > 110 ms, abnormal electrical axis, PR interval > 220 ms and conduction abnormalities) considered clinically significant by the investigator
* History of cardiac arrhythmias, ischemic heart disease or cerebrovascular disease
* Lower spinal malformation on physical or lumbar spine radiography, local spinal infection, or other abnormality, including but not limited to obesity, that would prevent LP or insertion of an indwelling catheter for CSF sampling
* Any history of seizure disorder, symptomatic seizures (not including a history of simple febrile seizures in childhood) or any past or present medical condition which, in the opinion of the investigator has the potential to reduce seizure threshold (e.g., history of head trauma or concussion, previous alcohol abuse, substance abuse).

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2012-07; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in cerebrospinal fluid amyloid-beta levels | baseline to 36 hours post-dose

SECONDARY OUTCOMES:
Incidence of adverse events | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Hakop Gevorkyan, Principal Investigator — California Clinical Trials Medical Group Inc.; Olukemi Olugemo, MD, Principal Investigator — PAREXEL International - EPCU Baltimore
Locations (2):
- United States (2):
  - Glendale, California
  - Baltimore, Maryland